CLINICAL TRIAL: NCT00624312
Title: A Prospective, Randomized, Double-Blinded Control Study of Procrit Versus Placebo to Determine Efficacy in Pre-Operative Patients Undergoing Major Surgical Oncology Operations
Brief Title: Procrit Versus Placebo to Determine Efficacy in Pre-Operative Major Surgical Oncology Operations
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: Ortho Biotech, Inc. (Industry)
Responsible Party: Principal Investigator, Robert C. Martin, Professor, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 07.0048
Record Dates: First submitted 2008-02-15; First posted 2008-02-27 (Estimated); Last update posted 2021-08-06 (Actual); Status verified 2013-09

CONDITIONS: Cancer
Keywords: Procrit; Erythropoietin; Patients undergoing major surgical oncology operations
MeSH Terms: conditions — Neoplasms | interventions — Epoetin Alfa

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Pre-operatively randomized to Procrit
  Interventions: Drug: Procrit
- 2 (Placebo Comparator): Pre-operatively randomized to placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Procrit — 10 days prior to surgery - injection of 60,000 IU of Procrit
  Day of surgery - injection of 60,000 IU of Procrit
  Other Names: Epoetin Alfa
  Arms: 1
Drug: Placebo — 10 days prior to surgery - injection with 60,000 IU of placebo
  Day of surgery - injection with 60,000 IU of placebo
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a two-dose regimen of Procrit prior to a major surgical oncology operation.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing a major surgical oncology procedure as defined below:

  * Pancreatectomy
  * Hepatectomy
  * Esophagectomy
  * Gastrectomy
  * Retroperitoneal Sarcoma Resection
* 18 years of age and older
* Hemoglobin level of ≥ 10g/dL to < 13g/dL, within 10 days of enrollment
* If female of child-bearing potential, negative pregnancy test within 14 days prior to surgery
* If subject is a sexually active male or a sexually active female of child- bearing potential, subject agrees to use a medically accepted form of contraception from the time of enrollment to completion of all follow-up study visits
* IRB-approved informed consent, signed by the subject or the subject's legally authorized representative ≥ 18 years of age

Exclusion Criteria:

* Pre-operative hemoglobin level ≥ 13g/dL or < 10g/dL
* Uncontrolled hypertension (defined as a systolic pressure ≥ 160 and/or a diastolic pressure ≥ 110)
* History of allergy to Procrit®
* Known hypersensitivity to mammalian cell-derived products or human albumin
* History of spontaneous venous thrombotic vascular events
* Anemia due to factors other than cancer,(e.g. iron deficiency, B12 deficiency)
* History of (within 12 months) deep venous thrombosis (DVT), pulmonary embolus (PE), or other venous thrombotic events. Prior superficial thrombophlebitis is not an exclusion criterion
* History of (within 6 months) uncontrolled cardiac arrhythmias, cerebrovascular accident (CVA), transient ischemic attack (TIA), acute coronary syndrome (ACS), or other arterial thrombosis. ACS includes Unstable Angina, Q wave Myocardial Infarction (QwMI), and non-Q wave myocardial infarction (NQMI)
* Currently receiving therapeutic or prophylactic anticoagulants for conditions other than planned surgery. The only exceptions are low dose aspirin (≤ 325 mg/day) or low dose anticoagulant to maintain patency of intravenous (IV) lines
* Patient is a candidate for autologous blood transfusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-02; Primary Completion 2010-01 (Estimated); Study Completion 2010-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients receiving transfusion. | One Year

CONTACTS AND LOCATIONS:
Overall Officials: Robert Martin, MD, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville, Louisville, Kentucky, United States